CLINICAL TRIAL: NCT04636957
Title: A Phase III, Multicenter, Randomized, Evaluator-blinded, Parallel-Group, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Ciprofloxacin 0.3% Plus Fluocinolone Acetonide 0.025% Otic Solution in the Treatment of Acute Otitis Externa (AOE)
Brief Title: A Phase III Study of Ciprofloxacin Plus Fluocinolone in Acute Otitis Externa (AOE)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZK- CIPRO+FLUO-201911
Record Dates: First submitted 2020-10-28; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Acute Otitis Externa
Keywords: ciprofloxacin; fluocinolone acetonide 0.025%; AOE
MeSH Terms: interventions — Ciprofloxacin; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ciprofloxacin 0.3% plus fluocinolone acetonide 0.025% (Experimental): Warm the otic solution by holding the vial in the hands for 1 to 2 minutes. Twist off the vial cap. Tilt the subjects' head to one side to keep the affected ear up. Instill the content of 1 vial in the ear (0.25mL). Gently pull the outer ear lobe upward and outward to allow the solution to flow into the ear canal. Keep the subjects' head tilted sideways for approximately 5 minutes to allow the drug time to penetrate the ear. Use twice daily (every 12±1h , morning and evening) for 7 consecutive days.
  Interventions: Drug: Ciprofloxacin-Fluocinolone Acetonide, 0.3%-0.025% Otic Solution
- ciprofloxacin 0.3% (Active Comparator): Warm the otic solution by holding the vial in the hands for 1 to 2 minutes. Twist off the vial cap. Tilt the subjects' head to one side to keep the affected ear up. Instill the content of 1 vial in the ear (0.25mL). Gently pull the outer ear lobe upward and outward to allow the solution to flow into the ear canal. Keep the subjects' head tilted sideways for approximately 5 minutes to allow the drug time to penetrate the ear. Use twice daily (every 12±1h, morning and evening) for 7 consecutive days
  Interventions: Drug: Ciprofloxacin 0.3% solution

INTERVENTIONS:
Drug: Ciprofloxacin-Fluocinolone Acetonide, 0.3%-0.025% Otic Solution — 0.25mL/vial, each vial contains 0.75mg of ciprofloxacin and 0.0625mg of fluocinolone acetonide.
  Arms: ciprofloxacin 0.3% plus fluocinolone acetonide 0.025%
Drug: Ciprofloxacin 0.3% solution — 0.4mL/vial, each vial contains 1.2mg ciprofloxacin
  Other Names: CETRAXAL OTICO®
  Arms: ciprofloxacin 0.3%

SUMMARY:
This is a phase Ⅲ, multicenter, randomized, evaluator-blinded, parallel-group, active-controlled study to assess the efficacy and safety of ciprofloxacin 0.3% plus fluocinolone acetonide 0.025% otic solution vs ciprofloxacin 0.3% otic solution in the treatment of AOE, and to assess the pharmacokinetic properties in 12 selected adult subjects. Eligible subjects will be randomized at 1:1 ration to either the treatment arm or control arm. All subject will receive 7 consecutive days of either ciprofloxacin 0.3% plus fluocinolone acetonide 0.025% otic solution or ciprofloxacin 0.3% otic solution alone. The main objectives are to assess the efficacy and safety of ciprofloxacin 0.3% plus fluocinolone acetonide 0.025% otic solution in the treatment of AOE, and to assess the plasma concentration of ciprofloxacin and fluocinolone acetonide after multiple doses of test drug in 12 adult subjects, and evaluate the PK parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with age of ≥3 years.
2. Subjects with clinical diagnosis of unilateral Acute Otitis Externa (AOE) within 21 days (3 weeks) prior to screening.
3. Subjects with graded II or III of AOE must experience each of symptoms or signs: as at least 2 for swelling (0-3 scale) and 1 for otorrhea (0-3 scale) and 2 for tenderness (0-3 scale).
4. Willingness to prevent water getting into the ear canal through end of the study (e.g. refrain from swimming, wear shower caps to cover the ears during showers).
5. For adult subjects, ability to fully understand the clinical trial and provide written informed consent. For subjects under the legal age (≥8 years and <18 of age) and capable of giving informed consent, informed consent form sign by both the subject and the parent/legal guardian. For subjects under 8 years of age, signed consent form from the parent/legal guardian.
6. For females of childbearing potential (including partners of male subjects), not planning a pregnancy during the study and agree to use adequate birth control methods (from screening until 28 days after the final dose).

Exclusion Criteria:

1. Subjects with bilateral AOE
2. Subjects who can't accept otoscopy (≤6 years of age) or oto-endoscope (>6 years of age).
3. Previous episode of AOE within 4 weeks prior to enrollment, or 2 or more episodes of AOE within 6 months prior to enrollment.
4. Tympanic membrane perforation (including tympanostomy tubes).
5. Known or suspected of fungal or viral ear infections, cholesteatoma, otitis media, malignant otitis externa, mastoiditis, seborrheic dermatitis, neurodermatitis in the external ear canal, ear trauma or other non-infectious suppurative ear diseases.
6. Known or suspected of hearing loss.
7. History of malignant tumors in the external ear canal, or currently receiving chemotherapy or radiotherapy.
8. Current diagnosis of diabetes mellitus, psoriasis, immunodeficiency or history of drug abuse.
9. Current diagnosis of cardiovascular, respiratory, urinary, gastrointestinal and neurological diseases which require intervention after at least 4 weeks of drug therapy.
10. Use of any systemic antibacterial or topical antibiotic, corticosteroids, analgesic and anti-inflammatory drugs and other drug that affect the study results within 1 week prior to screening.
11. Known or suspected hypersensitivity to quinolones, corticosteroid or any component of the study medication.
12. Participation in another clinical trial within the previous 3 months.
13. Pregnant women or nursing mothers.
14. Any condition that, in the judgment of the principal investigator, render the subject not suitable for the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 15 days after first dose
  The proportion of patients who have all symptoms scored as 0. Treatment failure is defined as any symptoms scored > 0.
  1. Swelling:
     None(0), Mild(1), Moderate(2), Severe(3).
  2. Otorrhea:
     None(0), Mild(1), Moderate(2), Severe(3).
  3. Tenderness:
  None(0), Mild(1), Moderate(2), Severe(3).

SECONDARY OUTCOMES:
Microbiological cure | 8 and 15 days after first dose
  Microbiological response will be classified as Eradicated, Presumed Eradicated, Persistence, Presumed Persistence, Partial Eradication, Superinfection and Reinfection. Microbiological cure rate is defined as the percentage of patients who achieve the eradication and presume eradication.
Overall therapeutic cure | 8 and 15 days after first dose
  Overall therapeutic cure will only be assessed among subjects whose microbiological culture are positive at baseline. Overall therapeutic cure is defined as the percentage of patients who achieve both clinical cure and microbiological cure.
Clinical cure | 8 days after first dose
  same as primary outcome measure
Change in clinical improvement | 8 and 15 days after first dose
  The percentage of patients whose any symptoms (swelling, otorrhea, tenderness) is improved ≥1 grade, compared to the first day
change in each of Signs and Symptoms | 8 and 15 days after first dose
  The percentage of patients whose each of signs and symptoms (swelling, otorrhea or tenderness) is improved ≥1 grade, compared to the first day
Change in Granulation Tissue | 8 and 15 days after first dose
  Granulation tissue will be scored as either 1=present or 0=absent. Improve rate of granulation tissue is defined as the percentage of patients whose granulation tissue in external ear canal at baseline is absent on 8 and 15 days after first dose
Change in ear pain | 8 and 15 days after first dose
  Pain improvement is defined as ear pain improved ≥1 grade on 8 and 15 days after first dose, compared to the first day.
Time to end of ear pain | 8 and 15 days after first dose
  Time to end of ear pain is the interval (in days) between the first dose of the study medication and the day of the cessation of the ear pain in the evaluable ear and will not recur until the end of the study. Time to end of ear pain in the whole group.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & Ent Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No